## Effect of Professional Prophylaxis on Clinical Parameters and Patient Comfort:Randomized Split-Mouth Clinical Trial

CONSENT TO PARTICIPATION



Researcher:

Signature

## CONSENT TO PARTICIPATION

**STUDY:** Comparison of the effect of prophylactic techniques in oral hygiene consultations on periodontal parameters and patient satisfaction.

| Oral Hygienist Telm: |
|---|
| The aim of this study is to compare professional oral health prophylaxis protocols. Participation in the study is voluntary and free of charge. |
| Procedures: If you agree to participate in this study, we will ask you to do the following: |
| <ul> <li>Answer a questionnaire in the form of an interview (5 minutes).</li> <li>The questionnaire has questions that aim to characterize sociodemographics, the general state of health as well as the care they usually have with the mouth.</li> <li>Allow a clinical observation of the teeth and gums to take about 20 minutes.</li> <li>For this observation, a mouth mirror and an instrument called a periodontal probe will be used to assess the health of the gums. Oral hygiene of the teeth will also be evaluated.</li> <li>These procedures are pain-free and not experimental, and they do not present any risks beyond those expected in any routine examination.</li> <li>Allow you to have an oral hygiene consultation using two different techniques.</li> <li>These procedures are pain-free and not experimental, will be performed by an experienced and trained professional and do not present any risks beyond those expected in any oral hygiene consultation.</li> <li>Answer a written questionnaire (2 minutes) about the satisfaction of the procedures performed.</li> <li>Allow two clinical observations to be made to the teeth and gums later, which will take about 20 minutes.</li> </ul> |
| <b>Additional information:</b> Your identification will never be disclosed and the information provided and collected is confidential, and is only available to researchers. You can ask as many questions as you want whenever you want. You can change your mind and to give up participating, at any time and without any consequence, everything they have to do is to communicate to the investigator. |
| Investigator's Signature Date |
| Participant/Legal Representative Statement: The study was explained to me and I agree to participate in this activity. I was given the opportunity to ask questions, change your mind about participating in the study I know that I can withdraw by simply informing any of the people listed with this work. |
| Participant's Name: |